CLINICAL TRIAL: NCT01638897
Title: DF4 Connector System Post-Approval Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: DF4
Record Dates: First submitted 2012-07-03; First posted 2012-07-12 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Sudden Cardiac Death; Heart Failure
Keywords: ICD; CRTD; DF4
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate long-term performance of the DF4 Connector System. This evaluation is based on the number of DF4 lead-related complications occurring during the study compared to the number of leads enrolled in the study. The DF4 systems will be followed for 5 years after implant. This study is required by FDA as a condition of approval of the DF4 Connector Systems. This study is conducted within Medtronic's post-market surveillance platform.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Subject is intended to be implanted or is within 30 days post-implant of a DF4 Connector System with a Medtronic DF4 lead used for a pacing, sensing and/or defibrillation application

Exclusion Criteria:

* Subject who is, or will be inaccessible for follow-up at a study site
* Subject with exclusion criteria required by local law (Europe, Central Asia [ECA] only)
* Implant and follow-up data, including any adverse device effects and system modifications at implant through the time of enrollment are unavailable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients intended to be implanted or are within 30 days post-implant of a DF4 Connector System with a Medtronic DF4 lead. All subjects must meet Inclusion criteria and none of the Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1778 (Actual)
Dates: Start 2012-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
DF4 Lead Related Complication Rate | Up to 5 Years
  To demonstrate that the complication-free probability is greater than 92.5% at five years post-implant for the high voltage DF4 lead

SECONDARY OUTCOMES:
Types of DF4 lead related events | Up to 5 years
  Number of DF4 lead related events grouped by type
Bipolar pacing impedance (ohms) | 5 years
  Summary statistics at 5 years post-implant will be reported.
High voltage impedance (ohms) | 5 years
  Summary statistics at 5 years post-implant will be reported
Pacing threshold (volts) | 5 years
  The pacing threshold is the minimum electrical stimulus needed to consistently depolarize the heart outside of the heart's refractory period. Summary statistics at 5 years post-implant will be reported.
Sensing amplitude (millivolts) | 5 years
  The amplitude of the intrinsic cardiac electrical signals detected by electrodes on the defibrillator lead will be summarized at 5 years post-implant.

CONTACTS AND LOCATIONS:
Locations (78):
- United States (72):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Gilbert, Arizona
  - Scottsdale, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - Rancho Mirage, California
  - Salinas, California
  - San Diego, California
  - San Francisco, California
  - Torrance, California
  - Van Nuys, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Albany, Georgia
  - Atlanta, Georgia
  - Marietta, Georgia
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Hyattsville, Maryland
  - Takoma Park, Maryland
  - Worcester, Massachusetts
  - Lansing, Michigan
  - Marquette, Michigan
  - Robbinsdale, Minnesota
  - Saint Louis Park, Minnesota
  - Saint Paul, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Henderson, Nevada
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - Garden City, New York
  - Huntington, New York
  - New York, New York
  - Poughkeepsie, New York
  - Utica, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Allentown, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Plano, Texas
  - The Woodlands, Texas
  - Burlington, Vermont
  - Olympia, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (5):
  - Calgary, Alberta
  - Kingston, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Trois-Rivières, Quebec
- Nantes, France